CLINICAL TRIAL: NCT01057225
Title: A Phase I/II Trial of Cyclophosphamide, Carfilzomib, Thalidomide and Dexamethasone (CYCLONE) in Patients With Newly Diagnosed Active Multiple Myeloma
Brief Title: Cyclophosphamide, Carfilzomib, Thalidomide, and Dexamethasone in Treating Patients With Newly Diagnosed Active Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0982; NCI-2009-01699 (Registry Identifier: NCI-CTRP); PT-171-502 (Other: Onyx Protocol); 09-004091 (Other: Mayo Clinic IRB); MC0982 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Results first posted 2016-09-23 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Cyclophosphamide; Thalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive carfilzomib IV on days 1, 2, 8, 9, 15, and 16; oral cyclophosphamide on days 1, 8, and 15; oral dexamethasone on days 1, 8, 15, and 22; and oral thalidomide on days 1-28.
  Interventions: Drug: carfilzomib; Drug: cyclophosphamide; Drug: thalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: carfilzomib — Given IV
  Other Names: PR-171
Drug: cyclophosphamide — Given orally
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Drug: thalidomide — Given orally
  Other Names: alpha-phthalimidoglutarimide; Contergan; Kevadon; Synovir; THAL; Thalomid
Drug: dexamethasone — Given orally
  Other Names: Aeroseb-Dex; Decaderm; Decadron; Decaspray; DM; DXM

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Thalidomide may stop the growth of cancer cells by blocking blood flow to the tumor. Giving combination chemotherapy together with carfilzomib and thalidomide may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of carfilzomib when given together with cyclophosphamide, thalidomide, and dexamethasone in treating patients with newly diagnosed active multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose of carfilzomib given in combination with oral cyclophosphamide and thalidomide and dexamethasone. (Phase I) II. In newly diagnosed myeloma to evaluate the response rate (CR, nCR, and VGPR) to carfilzomib given in combination with oral cyclophosphamide and thalidomide and dexamethasone after four 28 day cycles. (Phase II)

SECONDARY OBJECTIVES:

I. Determine the overall response rate (CR, nCR, PR) after 4, 8, 12 cycles. II. Determine the duration of progression-free and overall survival for patients receiving this regimen.

III. To evaluate the incidence of toxicities for this regimen. IV. To evaluate the ability to successfully collect peripheral blood stem cells following four months of combination therapy.

OUTLINE: This is a phase I, dose escalation study of carfilzomib followed by a phase II study.

Patients receive carfilzomib IV on days 1, 2, 8, 9, 15, and 16; oral cyclophosphamide on days 1, 8, and 15; oral dexamethasone on days 1, 8, 15, and 22; and oral thalidomide on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 3 months, then every 3 months for 1 year, and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion

* Creatinine =< 2 mg/dL
* Calculated Creatinine Clearance >= 30 mL/min
* Total Bilirubin =< 2.0 mg/dL
* Alkaline Phosphatase =< 3 x ULN
* ALT =< 3 x ULN
* Absolute neutrophil count >= 1000/uL
* Platelet >= 75000/uL
* Hemoglobin >= 8.0 g/dL
* Untreated symptomatic myeloma: Prior non-systemic therapy for the treatment of solitary plasmacytoma is permitted, but >= 1 month should have elapsed from the last day of radiation; prior therapy with clarithromycin, DHEA, anakinra, pamidronate or zoledronic acid is permitted; any additional agents not listed must be approved by the Principal Investigator
* Prior high dose corticosteroid therapy for twelve days (480 mg total dose) or less is permitted for emergent complications from newly diagnosed multiple myeloma
* Measurable disease of multiple myeloma, as defined by at least ONE of the following:
* Serum monoclonal protein >= 1.0 g by protein electrophoresis
* OR > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
* OR serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio; OR monoclonal bone marrow plasmacytosis >= 30% (evaluable disease)
* ECOG performance status (PS) 0, 1, 2; ECOG PS of 3 will be allowed if secondary to pain in the opinion of the Investigator
* Willingness and able to provide informed written consent
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willingness to return to Mayo Clinic enrolling institution for follow-up

Exclusion

* MGUS or smoldering myeloma
* Peripheral sensory neuropathy >= Grade 2 as defined by CTEP Active Version of the CTCAE
* Active malignancy with the exception of non melanoma skin cancer or in situ cervical or breast cancer
* Pregnant women or women of reproductive ability who are unwilling to use effective contraception
* Nursing women
* Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment
* Known hypersensitivity, allergy or inability to tolerate any of the agents employed
* Active, uncontrolled infection
* Severe cardiac comorbidity
* New York Heart Association Class III or IV Heart Failure
* Recent history of myocardial infarction in the six months prior to registration
* Uncontrolled angina or electrocardiographic evidence of acute ischemia
* Severe uncontrolled ventricular arrhythmias or electrocardiographic evidence of active conduction system abnormalities
* Cardiac amyloidosis with hypotension (systolic BP less than 100 mmHg)
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* The following medications are not permitted during the trial: any other investigational treatment; any cytotoxic chemotherapy; any other systemic anti-neoplastic therapy including, but not limited to, immunotherapy, hormonal therapy, or monoclonal antibody therapy
* Palliative radiation therapy is permitted if clinically indicated and not indicative of progressive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2017-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R. Mikhael, M.D., Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Level -1: Patients receive:
  Oral 300 mg/m^2 cyclophosphamide on days 1, 8, and 15;
  Oral 40 mg dexamethasone on days 1, 8, 15, and 22;
  Oral 100 mg thalidomide on days 1-28.
  Patients also recieve 15 mg/m^2 carfilzomib IV on days 1, 2, 8, 9, 15, and 16 in cycle 1, and 20 mg/m^2 on days 1, 2, 8, 9, 15, and 16 in subsequent cycles.
- Phase I: Dose Level 0; Phase II: Dose Level 0: Patients receive:
  Oral 300 mg/m^2 cyclophosphamide on days 1, 8, and 15;
  Oral 40 mg dexamethasone on days 1, 8, 15, and 22;
  Oral 100 mg thalidomide on days 1-28.
  Patients also recieve 20 mg/m^2 carfilzomib IV on days 1, 2, 8, 9, 15, and 16 in cycle 1, and 27 mg/m^2 on days 1, 2, 8, 9, 15, and 16 in subsequent cycles.
- Phase I: Dose Level 1; Phase II: Dose Level 1: Patients receive:
  Oral 300 mg/m^2 cyclophosphamide on days 1, 8, and 15;
  Oral 40 mg dexamethasone on days 1, 8, 15, and 22;
  Oral 100 mg thalidomide on days 1-28.
  Patients also recieve 20 mg/m^2 carfilzomib IV on days 1, 2, 8, 9, 15, and 16 in cycle 1, and 36 mg/m^2 on days 1, 2, 8, 9, 15, and 16 in subsequent cycles.
- Phase I: Dose Level 2: Patients receive:
  Oral 300 mg/m^2 cyclophosphamide on days 1, 8, and 15;
  Oral 40 mg dexamethasone on days 1, 8, 15, and 22;
  Oral 100 mg thalidomide on days 1-28.
  Patients also recieve 20 mg/m^2 carfilzomib IV on days 1, 2, 8, 9, 15, and 16 in cycle 1, and 45 mg/m^2 on days 1, 2, 8, 9, 15, and 16 in subsequent cycles.
Period: Overall Study
Arm/Group | Phase I: Dose Level -1 | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II: Dose Level 0 | Phase II: Dose Level 1
Started | 3 | 3 | 6 | 7 | 22 | 23
Completed | 3 | 3 | 6 | 7 | 22 | 23
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that were eligible and treated for the study were evaluated.
Groups:
- All Treated Patients: Patients receive carfilzomib IV on days 1, 2, 8, 9, 15, and 16; oral cyclophosphamide on days 1, 8, and 15; oral dexamethasone on days 1, 8, 15, and 22; and oral thalidomide on days 1-28.
Arm/Group | All Treated Patients
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 62.5 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 54
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (Phase I)
Description: To establish the maximum tolerated dose of carfilzomib given in combination with oral cyclophosphamide and thalidomide and dexamethasone.
  For this protocol, dose-limiting toxicity (DLT) will be defined as an adverse event attributed (definitely, probably, possibly) in the first or second cycle for patients enrolled to Dose Levels -1 and 0 and in the first cycle only for patients enrolled to Dose Levels 1 and 2.
  We are reporting the number of DLTs
Time Frame: From baseline to end of active treatment, up to 12 28-day cycles.
Population: All patients registered to a dose escalation Phase I group were analyzed for this endpoint.
Measure: Number; unit: participants
Arm/Group | Phase I: Dose Level -1 | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2
Number analyzed (Participants) | 3 | 3 | 6 | 7
participants | 0 | 0 | 0 | 3
Statistical Analysis 1: Comparison: Phase I: Dose Level -1 vs Phase I: Dose Level 0 vs Phase I: Dose Level 1 vs Phase I: Dose Level 2; Test type: Superiority or Other; Dose Level = 1 — Using a cohort of 3 design, it was determined the maximum tolerated dose of carfilzomib is Dose Level 1: 20 mg/m^2 for the first cycle and 36 mg/m^2 for subsequent cycles

2. Primary Outcome: Percentage of Patients Who Have at Least a Confirmed Very Good Partial Response (Phase II)
Description: The proportion of patients who have at least a confirmed very good partial response will be calculated by taking the number of patients with a very good partial response or a complete response divided by the total number of patients.
  A complete response is defined as:
  * Negative immunofixation of the serum and urine
  * If at on study, only the measurable non-bone marrow parameter was FLC, normalization of FLC ratio
  * < 5% plasma cells in bone marrow
  * Disappearance of any soft tissue plasmacytomas
  A very good partial response is defined as:
  * Serum and urine M-component detectable by immunofixation but not on electrophoresis or
  * If at on study, serum measurable, ≥ 90% or greater reduction in serum Mcomponent
  * Urine M-component <100 mg per 24 hour
Time Frame: Following the first 4 cycles of treatment (28 day cycles)
Population: All enrolled patients who began treatment were evaluated for safety and response.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 64
percentage of participants | 91

3. Secondary Outcome: Progression-free Survival (Phase II)
Description: PFS was defined as the time from registration to progression or death due to any cause. Progression was defined as any one or more of the following:
  • Increase of 25% from lowest confirmed response in: Serum M-component (absolute increase must be ≥ 0.5 g/dl)c Urine M-component (absolute increase must be ≥ 200 mg/24 hour) If at on study, only the measurable non-bone marrow parameter was FLC, the difference between involved and uninvolved FLC levels (absolute increase must be >10 mg/dl) Bone marrow plasma cell percentage (absolute % must be 10%)d Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
  • Development of hypercalcemia (corrected serum calcium >11.5 mg/dl) that can be attributed solely to the plasma cell proliferative disorder
Time Frame: From baseline to progression or death up to 3 years
Population: All of the 64 participants that were eligible and began treatment were evaluated.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 64
months | NA [NA to NA] — The median and 95% confidence interval for the progression free survival could not be estimated due to too few events.

4. Secondary Outcome: Time to Treatment Failure
Description: The time from the date of registration to the date at which the patient is removed from treatment due to progression, adverse events, or refusal. If the patient is considered to be a major treatment violation or is taken off study as a non-protocol failure, the patient will be censored on the date they were removed from treatment. The distribution of time to treatment failure will be estimated using the method of Kaplan-Meier
Time Frame: From baseline to end of active treatment
Population: All enrolled patients who began treatment were evaluated for safety and response.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 64
months | NA [NA to NA] — The median and 95% confidence interval for the time to treatment failure could not be estimated due to too few treatment failures.

5. Secondary Outcome: Stem Cell Collection and Engraftment (Phase II)
Description: For patients going on to stem cell collection, the total number of CD34 positive cells collected per collection, days to platelets over 20,000 without transfusion and ANC over 1000 will be recorded. If a patient fails to collect adequate stem cells for transplant, this will be recorded as such. The number of patients with successful stem cell mobilization are reported.
Time Frame: Following the first 4 courses of treatment
Population: Of the 64 patients that began protocol treatment, stem cell harvesting was attempted on 42 patients.
Measure: Number; unit: participants
Arm/Group | All Treated Patients
Number analyzed (Participants) | 42
participants | 42

6. Secondary Outcome: Complete Response (Phase II)
Description: In patients continuing beyond 4 cycles the ability to induce complete response will be evaluated at completion of planned therapy.
Time Frame: Following the first 4 courses of treatment
Measure: Number; unit: participants
Groups:
- Dose Level -1: Patients receive:
  Oral 300 mg/m^2 cyclophosphamide on days 1, 8, and 15;
  Oral 40 mg dexamethasone on days 1, 8, 15, and 22;
  Oral 100 mg thalidomide on days 1-28.
  Patients also recieve 15 mg/m^2 carfilzomib IV on days 1, 2, 8, 9, 15, and 16 in cycle 1, and 20 mg/m^2 on days 1, 2, 8, 9, 15, and 16 in subsequent cycles.
- Dose Level 0: Patients receive:
  Oral 300 mg/m^2 cyclophosphamide on days 1, 8, and 15;
  Oral 40 mg dexamethasone on days 1, 8, 15, and 22;
  Oral 100 mg thalidomide on days 1-28.
  Patients also recieve 20 mg/m^2 carfilzomib IV on days 1, 2, 8, 9, 15, and 16 in cycle 1, and 27 mg/m^2 on days 1, 2, 8, 9, 15, and 16 in subsequent cycles.
- Dose Level 1: Patients receive:
  Oral 300 mg/m^2 cyclophosphamide on days 1, 8, and 15;
  Oral 40 mg dexamethasone on days 1, 8, 15, and 22;
  Oral 100 mg thalidomide on days 1-28.
  Patients also recieve 20 mg/m^2 carfilzomib IV on days 1, 2, 8, 9, 15, and 16 in cycle 1, and 36 mg/m^2 on days 1, 2, 8, 9, 15, and 16 in subsequent cycles.
- Dose Level 2: Patients receive:
  Oral 300 mg/m^2 cyclophosphamide on days 1, 8, and 15;
  Oral 40 mg dexamethasone on days 1, 8, 15, and 22;
  Oral 100 mg thalidomide on days 1-28.
  Patients also recieve 20 mg/m^2 carfilzomib IV on days 1, 2, 8, 9, 15, and 16 in cycle 1, and 45 mg/m^2 on days 1, 2, 8, 9, 15, and 16 in subsequent cycles.
Arm/Group | Dose Level -1 | Dose Level 0 | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 3 | 25 | 29 | 7
participants | 0 | 2 | 3 | 0

7. Secondary Outcome: Survival Time (Phase II)
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier
Time Frame: From baseline to death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Treated Patients
Number analyzed (Participants) | 64
months | NA [NA to NA] — The median and 95% confidence interval for the survival time could not be estimated due to too few deaths.

8. Secondary Outcome: Progression Free Survival (12 Month)
Description: Progression-free survival time is defined as the time from registration to the earliest date of documentation of disease progression. If a patient dies without a documentation of disease progression the patient will be considered to have had disease progression at the time of their death. If the patient is declared to be a major treatment violation, the patient will be censored on the date the treatment violation was declared to have occurred. In the case of a patient starting treatment and then never returning for any evaluations, the patient will be censored for progression 1 day post-registration. This is reported as the percentage of patients alive and progression free at the 12 month mark.
Time Frame: 12 months
Population: All of the 64 participants that were eligible and began treatment were evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of participants at 12 months
Arm/Group | All Treated Patients
Number analyzed (Participants) | 64
percentage of participants at 12 months | 85 [71 to 93]

9. Secondary Outcome: Progession Free Survival (24 Month)
Description: Progression-free survival time is defined as the time from registration to the earliest date of documentation of disease progression. If a patient dies without a documentation of disease progression the patient will be considered to have had disease progression at the time of their death. If the patient is declared to be a major treatment violation, the patient will be censored on the date the treatment violation was declared to have occurred. In the case of a patient starting treatment and then never returning for any evaluations, the patient will be censored for progression 1 day post-registration. This is reported as the percentage of patients alive and progression free at the 24 month mark.
Time Frame: 24 months
Population: All of the 64 participants that were eligible and began treatment were evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of participants at 24 months
Arm/Group | All Treated Patients
Number analyzed (Participants) | 64
percentage of participants at 24 months | 76 [59 to 87]

10. Secondary Outcome: Overall Survival (12 Month)
Description: 12 Month Overall survival is defined as the proportion of patients to still be alive after 12 months.
Time Frame: From baseline to death
Population: All of the 64 participants that were eligible and began treatment were evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | All Treated Patients
Number analyzed (Participants) | 64
percentage of patients | 96 [86 to 99]

11. Secondary Outcome: Overall Survival (24 Month)
Description: 24 Month Overall survival is defined as the proportion of patients to still be alive after 24 months.
Time Frame: From baseline to death
Population: All of the 64 participants that were eligible and began treatment were evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | All Treated Patients
Number analyzed (Participants) | 64
percentage of patients | 96 [86 to 99]

ADVERSE EVENTS:
Arm/Group | All Treated Patients
Serious Adverse Events (participants affected / at risk) | 30/64
Other Adverse Events (participants affected / at risk) | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Patients (N=64)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (2)
Heart failure (Cardiac disorders) | 3 (3)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Infusion related reaction (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 4 (4)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Creatinine increased (Investigations) | 3 (4)
Lymphocyte count decreased (Investigations) | 2 (5)
Neutrophil count decreased (Investigations) | 3 (3)
Urine output decreased (Investigations) | 1 (4)
White blood cell decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 4 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Patients (N=64)
Anemia (Blood and lymphatic system disorders) | 27 (74)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (4)
Cushingoid (Endocrine disorders) | 1 (2)
Floaters (Eye disorders) | 1 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Constipation (Gastrointestinal disorders) | 35 (106)
Diarrhea (Gastrointestinal disorders) | 10 (17)
Dry mouth (Gastrointestinal disorders) | 2 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (5)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (22)
Vomiting (Gastrointestinal disorders) | 3 (4)
Chills (General disorders) | 3 (3)
Edema limbs (General disorders) | 15 (28)
Edema trunk (General disorders) | 2 (2)
Fatigue (General disorders) | 51 (159)
Fever (General disorders) | 5 (5)
Gait disturbance (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (2)
Irritability (General disorders) | 2 (4)
Malaise (General disorders) | 11 (34)
Pain (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 7 (12)
Alkaline phosphatase increased (Investigations) | 9 (12)
Aspartate aminotransferase increased (Investigations) | 8 (13)
Blood bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 24 (54)
Investigations - Other, specify (Investigations) | 2 (5)
Lymphocyte count decreased (Investigations) | 26 (112)
Lymphocyte count increased (Investigations) | 4 (5)
Neutrophil count decreased (Investigations) | 32 (95)
Platelet count decreased (Investigations) | 30 (74)
Weight gain (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 27 (76)
Anorexia (Metabolism and nutrition disorders) | 6 (9)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 24 (79)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (7)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 14 (30)
Hypokalemia (Metabolism and nutrition disorders) | 10 (22)
Hyponatremia (Metabolism and nutrition disorders) | 9 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (14)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 7 (8)
Dizziness (Nervous system disorders) | 7 (12)
Dysgeusia (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 7 (13)
Lethargy (Nervous system disorders) | 16 (22)
Memory impairment (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (3)
Peripheral motor neuropathy (Nervous system disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 23 (65)
Seizure (Nervous system disorders) | 1 (3)
Somnolence (Nervous system disorders) | 13 (19)
Tremor (Nervous system disorders) | 4 (11)
Anxiety (Psychiatric disorders) | 5 (10)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (4)
Insomnia (Psychiatric disorders) | 4 (5)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (4)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (2)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (21)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (8)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (4)
Hypertension (Vascular disorders) | 5 (19)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes